CLINICAL TRIAL: NCT02163395
Title: A Prospective Open Label Single Arm Study to Evaluate the Performance of Straumann Monotype FullCeram (Zirconium Dioxide) Implants in Single Tooth Gaps in the Maxilla and Mandible
Brief Title: Performance Evaluation of FullCeram Implants in Single Tooth Gaps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR 01/07
Record Dates: First submitted 2014-06-10; First posted 2014-06-13 (Estimated); Results first posted 2015-07-16 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2022-05

CONDITIONS: Tooth Loss
Keywords: Ceramic implant
MeSH Terms: conditions — Tooth Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FullCeram implant (Other): Straumann FullCeram Implant is a monotype ZrO2 implant with a diameter of 4.1 mm, available in lengths of 8, 10, 12 and 14 mm and abutment heights of 4.0 or 5.5 mm
  Interventions: Device: FullCeram implant

INTERVENTIONS:
Device: FullCeram implant — FullCeram implantation
  Other Names: Straumann Monotype FullCeram (Zirconium dioxide)

SUMMARY:
* Straumann Monotype FullCeram implants serve as a suitable alternative for implant therapy especially in the aesthetic zone
* The survival rate of Straumann Ceramic implants should be at least 85% (max 6 implant losses out of 40 patients) after the first year

DETAILED DESCRIPTION:
This is a prospective, open label, single arm, multicenter study. The total study duration for each patient was prolonged to 10 years follow-up. It is acceptable to have the visit performed up to 6 month after the aspired date.

The primary study parameter will be analyzed as soon as every patient passed visit 6 (annual follow-up visit, 12 month +/- 4 weeks).

Implants will be placed transmucosally and will be protected by a thermoplastic splint for healing. A provisional prosthesis will be placed (out of occlusion) 12-14 weeks post implant placement. The final crown will be done between study week 24 and 28. Implant survival, implant success, bone loss, periodontal parameters and adverse events will be assessed in the follow-up visits.

In total 10 visits are scheduled in this study. The investigational device: Straumann FullCeram Implant is a monotype ZrO2 implant with a diameter of 4.1 mm, available in lengths of 8, 10, 12 and 14 mm and abutment heights of 4.0 or 5.5 mm. This is a CE marked product.

Three centres in Germany are participating. The study and any amendments will be performed as far as possible according to ISO 14155 (Second Edition, 2011-02-01) and conform to the Declaration of Helsinki (last revised Seoul 2008) and local legal and regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have voluntary signed the informed consent and the data protection consent form before any study related action
* Males and females with at least 18 years of age (including 18 years)
* Implant placement planned in the maxilla or mandible
* The missing tooth site must have a tooth with a natural root
* Substantially healed and augmented extraction sockets (minimal 8 weeks)
* Autogenous bone augmentation until 3 month pre-implantation were bone deficiency jeopardizing the implant position

Exclusion Criteria:

Pre-surgical exclusion criteria:

* Systemic disease that would interfere with dental implant therapy
* Any contraindications for oral surgical procedures
* Mucosal diseases
* History of local irradiation therapy
* Current untreated periodontitis or gingivitis
* Any untreated endodontic lesions
* Probing pocket depth of > or = 4 mm on one of the teeth immediately adjacent to the dental implant site
* Severe bruxing or clenching habits
* Patients with inadequate oral hygiene or unmotivated for adequate home care
* Patients who smoke >10 cigarettes per day or tobacco equivalents or chew tobacco
* Subjects who have undergone administration of any investigational device within 30 days of enrolment in the study
* Conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance or unreliability
* Physical or mental handicaps that would interfere with the ability to perform adequate oral hygiene
* Pregnant women at screening

Secondary exclusion criteria at or after implant surgery:

* Lack of primary stability of the implant (hand testing directly after surgery)
* Inappropriate implant position for the prosthetic requirements (to be estimated before provisional restoration)
* Major simultaneous augmentation procedures (at surgery)
* X-ray of implant does not show the implant from first bone contact to apical tip (at surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2023-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gahlert, Prof Dr Dr, Principal Investigator — Oralchirurgie T1
Locations (3):
- Germany (3):
  - Medizinische Hochschule Hannover Klinik und Poliklinik fuer Mund-, Kiefer- und Gesichtschirurgie, Hanover
  - Oralchirurgie T1, Munich
  - Katharinenhospital, Stuttgart

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lambrecht TJ, Filipi A, Raetzer Luenzel A, Schiel HJ. Long-Term evaluation of submerged and nonsubmerged ITI solid-screw titanium implants. A 10-year life table analysis of 468 implants. Int J Oral Maxifollofac Implants; 18:826-834, 2003. Kohal R J, et al. Loaded custom-made zirconia and titanium implants show similar osseointegration: an animal experiment. J Periodontol. 75.9, 1262-68, 2004. Scarano A, et al. Bone response to zirconia ceramic implants: an experimental study in rabbits. J Oral Implantol. 8-12, 29.1, 2003. Sennerby L, at al. Bone tissue resonses to surface-modified zirconia implants: A histomorphometric and removal torque study in the rabbit. Clin. Implant. Dent.Relat Res. 7 Suppl: S13-S20, 2005. Blaschke C, and Volz U. Soft and hard tissue response to zirconium dioxide dental implants - a clinical study in man. Neuro.Endocrinol.Lett. 27.Suppl1, 2006. Olivia J, Olivia X, Olivia JD. One year follow-up of first consecutive 100 Zirconia Dental Implants in humans: A comparison of 2 different rough surfaces. Int J Oral Maxillofac Implants; 22:430-435, 2007. Herrmann JS, Buser D, Schenk RK, Schoolfield JD, Cochran DL. Biologic width around one-and two-piece titanium implants. A histometric evaluation of unloaded nonsubmerged and submerged implants in the canine mandible. Clin Oral Impl Res 12, 559-571, 2001. Todescan FF, Pustiglioni FE, Imbronito AV, Albrektson T, Gioso M. Influenze of the microgap in the peri-implant hard and soft tissues. A histomorphometric study in dogs. Int J Pral Maxillofac Implants 17:467-472, 2002. Buser D, Weber HP, Braegger U, Balsinger C. Gewebeintegration einphasiger ITI-Implantate: Drei-Jahres-Ergebnisse einer prospektiven Langzeitstudie mit Hohlzylinder- und Hohlschraubenimplantaten. Buser D, Martin W, Belser UC. Optimizing Esthetics for Implant restorations in the Anterior Maxilla: Anatomic and Surgical Considerations. Int. J Oral and Maxillofacial Implants. Supplement; 19:43-61, 2004.
- [Derived] Bormann KH, Gellrich NC, Kniha H, Schild S, Weingart D, Gahlert M. A prospective clinical study to evaluate the performance of zirconium dioxide dental implants in single-tooth edentulous area: 3-year follow-up. BMC Oral Health. 2018 Nov 1;18(1):181. doi: 10.1186/s12903-018-0636-x. PMID 30382850

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FullCeram Implant
Started | 44
Completed | 39
Not Completed | 5
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 3
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | FullCeram Implant
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 17
Region of Enrollment [Number; unit: participants]
  Germany | 44

OUTCOME MEASURES:

1. Primary Outcome: The Implant Survival
Description: A surviving implant is an integrated implant in the patient's jaw bone at the time of assessment.
Time Frame: Measured at 12 months +/- 4 weeks after implant placement
Population: Implant survival rates provided for the patients of the ITT population, who had valid data. Missing data were not imputed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FullCeram Implant
Number analyzed (Participants) | 42
percentage of participants | 97.6 [86.6 to 99.9]

2. Secondary Outcome: The Implant Success
Description: According to Buser et al 1992 an implant will be deemed a success if all of the following success criteria apply.
  * Absence of persisting subjective discomfort such as pain, foreign body perception and or dysaesthesia (painful sensation)
  * Absence of a recurrent peri-implant infection with suppuration (where an infection is termed recurrent if it is observed at two or more follow-up visits after treatment with systemic antibiotics)
  * Absence of implant mobility on manual palpation
  * Absence of any continuous peri-implant radiolucency
Time Frame: Measured at Week 26, Month 12, Month 24 and Month 36
Population: Implant success rates provided for the patients of the ITT population, who had valid data. Missing data were not imputed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FullCeram Implant
Number analyzed (Participants) | 43
percentage of participants
  Week 26 (n=43) | 93.0 [80.7 to 98.3]
  Month 12 (n=42): number analyzed (Participants) | 42
  Month 12 (n=42) | 97.6 [86.6 to 99.9]
  Month 24 (n=41): number analyzed (Participants) | 41
  Month 24 (n=41) | 95.1 [83.0 to 99.5]
  Month 36 (n=40): number analyzed (Participants) | 40
  Month 36 (n=40) | 97.5 [86.0 to 99.9]

3. Secondary Outcome: Mean Bone Level Changes (Distal and Mesial)
Description: A radiographic stent was produced to have a standard measurement. The distal and mesial bone levels were combined into a single value by averaging the two values. Negative bone level changes representing bone loss between baseline and follow-up visits, vice versa positive changes representing bone gain.
Time Frame: Measured at Week 26, Month 12, Month 24 and Month 36
Population: Standardised bone level measurements provided for the ITT population. Missing data were not imputed.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | FullCeram Implant
Number analyzed (Participants) | 39
mm
  Week 26 (n=39) | -0.88 (0.86)
  Month 12 (n=39) | -1.02 (0.90)
  Month 24 (n=38): number analyzed (Participants) | 38
  Month 24 (n=38) | -1.24 (0.94)
  Month 36 (n=37): number analyzed (Participants) | 37
  Month 36 (n=37) | -0.97 (0.88)

4. Secondary Outcome: The Implant Survival
Description: A surviving implant is an integrated implant in the patient's jaw bone at the time of assessment.
Time Frame: Measured at Week 26, Month 24 and Month 36
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | FullCeram Implant
Number analyzed (Participants) | 43
percentage of participants
  Week 26 (n= 43) | 97.7 [86.6 to 99.9]
  Month 24 (n= 41): number analyzed (Participants) | 41
  Month 24 (n= 41) | 97.6 [86.3 to 99.9]
  Month 36 (n= 40): number analyzed (Participants) | 40
  Month 36 (n= 40) | 97.5 [86.0 to 99.9]

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were reported from the time a patient provided written informed consent to the 36-month follow-up visit.
Arm/Group | FullCeram Implant
Serious Adverse Events (participants affected / at risk) | 5/44
Other Adverse Events (participants affected / at risk) | 33/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FullCeram Implant (N=44)
Sepsis (Blood and lymphatic system disorders) | 1 (1) — not related
Fracture (Surgical and medical procedures) | 1 (1) — not related
Meniscus surgery (Musculoskeletal and connective tissue disorders) | 1 (1)
Birth of a boy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Hospitalization (General disorders) | 1 (1)
Calcaneal spur (Musculoskeletal and connective tissue disorders) | 1 (1)
Kidney infection (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FullCeram Implant (N=44)
Pain (General disorders) | 18 (18)
Bleeding, swelling, inflammation / infection (Surgical and medical procedures) | 10 (10)
Cold, influenza or sore throat (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Insufficient, loose or broken crown (Surgical and medical procedures) | 8 (8)
Implant success criteria not fulfilled (Surgical and medical procedures) | 3 (3)
Adenovirus (Infections and infestations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Decrease of gingiva (Skin and subcutaneous tissue disorders) | 1 (1)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pocket formation and bone loss (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Hypertonus (Cardiac disorders) | 1 (1)
Abdominal pain (General disorders) | 1 (1)
Accident (General disorders) | 1 (1)
Chronic bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic lymphocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid hypofunction (General disorders) | 1 (1)
Uterine abrasion (Reproductive system and breast disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No